CLINICAL TRIAL: NCT03721991
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Single-centre Trial of GABA Treatment in Subjects With Type 1 Diabetes
Brief Title: GABA Treatment in Subjects With Type 1 Diabetes
Acronym: GABA-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H17041847
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: beta cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: randomised controlled study with active compared to placebo for 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomised controlled with placebo tablets matching active capsules with investigational product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GABA (Active Comparator): gamma Amino butyric acid (GABA) food supplement with 6 g per day
  Interventions: Dietary Supplement: Gama amino butyric acid (GABA)
- PLACEBO (Placebo Comparator): Matching placebo capsules to GABA
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Gama amino butyric acid (GABA) — food supplement Gama amino butyric acid (GABA) as capsules
  Other Names: gaba
  Arms: GABA
Dietary Supplement: placebo — matching placebo
  Arms: PLACEBO

SUMMARY:
test if a food supplementation with GABA can improve insulin production capacity in type 1 diabetes patients by turning alfa cells into beta cells in accordance with mice and cell studies.randomised parallel study with placebo as control

DETAILED DESCRIPTION:
our results indicate that alfa-cells can be regenerated and used to regenerate functional beta-like cells in vivo in type 1 diabetes models. Aiming to eventually apply these findings to type 1 diabetic patients, we initiated multiple screens seeking for compounds inducing alfa-to-beta-cell conversion. Using the mouse as a model, we thereby found that GABA (gamma-aminobutyric acid) could promote a cycle of conversion of alfa-cells into functional beta-like cells,GABA being considered as a non-harmful food supplement, one could envision a trial in type 1 diabetic patients. Indeed, a putative cure for type 1 diabetes may include halting the autoimmune insult to the pancreatic beta-cells and restoring insulin secretion by expanding beta-cell mass by beta-cell-regeneration and/or preventing beta-cell apoptosis induced by cytokines. Immunosuppression initiated at the onset of type 1 diabetes has been shown to preserve beta-cell function, but is associated with significant toxicities. Other studies using nicotinamide and parenteral insulin have failed to prevent development of type 1 diabetes.

Objectives Primary objective: To investigate the effect and safety of the dietary supplement GABA provided at a dose of 6 g daily compared to placebo for 12 weeks on change in beta-cell function in patients with C-peptide negative type 1 diabetes as an adjunctive therapy to insulin treatment.

Population A total of 30 patients with C-peptide negative type 1 diabetes, randomised 2:1 GABA: Placebo.

Intervention After randomisation patients are treated with the dietary supplement GABA or matching placebo, titrated to 3 x 2g, or maximum tolerated dose, for 12 weeks. The insulin dose is reduced if needed according to Self-monitored blood glucose (SMBG) and hypoglycaemic episodes.

ELIGIBILITY:
Inclusion Criteria:stimulated c peptide <0.03 mmol/l type 1 diabetes

-

Exclusion Criteria:

* • Type 2 diabetes

  * Fertile women not using chemical (tablet/pill, depot injection of progesterone, subdermal gestagen implantation, hormonal vaginal ring or transdermal hormonal patch) or mechanical (spirals) contraceptives
  * Pregnant or nursing women
  * Cancer unless in complete remission for > 5 years
  * Treatment with oral glucocorticoids
  * Hypoglycaemia unawareness (unability to register low blood glucose)
  * Known or suspected hypersensitivity to trial product or related products
  * Abuse of alcohol or drugs, or any other co-existing condition that would make patients unsuitable to participate in the study, as deemed by the investigators
  * Receipt of an investigational drug within 30 days prior to visit 0
  * Simultaneous participation in any other clinical intervention trial
  * Chronic systemic use of steroids
  * Seizure disorder
  * Current use of Baclofen, Valium, Acamprosate, Neurontin, or Lyrica

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
insulin production | 12 weeks
  c peptide production during meal stimulation

SECONDARY OUTCOMES:
c peptide response (change from fasting baseline to meal stimulated concentration in blood) | after 12 weeks
  maximal c peptide change from baseline during meal testing with sustacal,
c peptide response beta cell | after 12 weeks
  beta cell sensitivity during meal testing, calculated with Homeostatic Model assessment b (HOMAb)
glucagon response | after 12 weeks
  increase in blood glucagon concentration from fasting to peak during meal testing,
metabolic parameters | 12 weeks
  hba1c (mmol/mol) change from baseline
metabolic parameters dose of insulin | 12 weeks
  insulin dose used pr 24 hours
metabolic parameters glucose | 12 weeks
  hypoglycemia,(number of events of severe and mild hypoglycemia self reported)
metabolic parameters lipid | 12 weeks
  lipid (LDL cholesterol ) (mmol/l)
metabolic parameters weight | 12 weeks
  body weight (kg)
metabolic parameters waist | 12 weeks
  waist circumference (cm)
metabolic parameters SMBG | 12 weeks
  SMBG self monitored blood glucose (mmol/l) 7 points profile in diary
metabolic parameters quality of life | 12 weeks
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: peter Rossing, md, Study Chair — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
data protection rules may not approve data sharing